CLINICAL TRIAL: NCT01757197
Title: Tocilizumab (an Anti-human IL-6 Receptor Monoclonal Antibody) as a First Line Therapy for Patients With Glucocorticoid-refractory Acute Graft vs. Host Disease (aGVHD) After Allogeneic Hematopoetic Stem Cell Transplant (HSCT), a Phase II Study.
Brief Title: Phase II Study of Tocilizumab for Patients With Glucocorticoid-refractory Acute GVHD After Allogeneic Hematopoetic Stem Cell Transplant (HSCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1202012180; ML28046 (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2012-12-13; First posted 2012-12-28 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Glucocorticosteroid Refractory Acute GVHD
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental): Toclizumab will be administered on Day 0. The administration of tocilizumab will be every 2 weeks for a total of 8 doses.
  Interventions: Drug: Toclizumab

INTERVENTIONS:
Drug: Toclizumab — 8 mg/kg IV, once every 1-2 weeks. The maximum dose per infusion should not exceed 800 mg.
  Other Names: ACTEMRA®

SUMMARY:
The purpose of this study is to determine if Tocilizumab is a safe and effective treatment for steroid-refractory acute graft versus host disease.

DETAILED DESCRIPTION:
This clinical trial is testing a drug called Tocilizumab (a monoclonal antibody) as a first line therapy for subjects with steroid-refractory acute graft versus host disease (acute GVHD) after undergoing a bone marrow transplant. The purpose of the study is to test the safety and efficacy of Tocilizumab at differing dose schedules. There are 2 phases to this study. Both phases include subjects with acute GVHD have not responded to steroid treatment. Subjects enrolled in Phase IIp will receive Tocilizumab 8 mg/kg every week or every 2 weeks. Subjects enrolled in Phase II will receive one of two dose schedules determined by the results of Phase IIp. Depending on the dose they are assigned to, subjects will receive Tocilizumab every week or every 2 weeks for a total of 8 doses. The study medication may be interrupted, withheld or stopped for different reasons. However, subjects will be asked to follow up periodically for one year after starting Tocilizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 80 years of age
* Karnofsky Performance Status Scale ≥ 50%
* Glucocorticosteroid refractory acute GVHD Grade 2-4 by the Glucksberg functional classification.
* Patients who had experienced aGVHD grade 2-4 and responded to glucocorticosteroids in the past then had a flare of aGVHD requiring increasing immune suppression to 1 mg/kg of prednisone or equivalent are eligible for this study if they are refractory to steroids and provided that they did not receive a second line therapy for aGVHD in the past.
* Glucocorticosteroid refractory GVHD is defined as the following:

  * No response to corticosteroid therapy at ≥ 1.0 mg/kg methylprednisolone or equivalent after the onset of acute GVHD for a minimum of 3 and a maximum of 7 days OR
  * Progression of at least 1 overall grade within 3 days of glucocorticosteroid use OR
  * Incomplete response by 14 days of glucocorticosteroid use
* Ability to comply with planned procedures
* Ability to understand the information provided and to provide written evidence of informed consent
* Willingness of females of childbearing potential to use adequate contraception.
* Post-menopausal for at least 1 year or surgical sterilization or hysterectomy at least 3 months prior to screening

Exclusion Criteria:

* Subjects with only grade 1 acute GVHD
* Concurrent medical condition or disease that may interfere with clinical trial participation
* Relapsed or persistent malignancy.
* Receiving other drugs for the treatment of glucocorticosteroid refractory GVHD.
* Severe hepatic veno-occlusive disease or sinusoidal obstruction syndrome.
* History of hypersensitivity or severe allergic reactions to humanized or murine monoclonal antibodies
* Receipt of any experimental, unregistered therapy within or outside a clinical trial within 30 days or 5 plasma half-lives (whichever is shorter) before dosing
* Planned or current participation in any other clinical trial for treatment of GVHD during this clinical trial. Subjects are permitted on this trial if 30 days (or 5 half-lives) have passed since enrollment on other investigational drugs. If a subject develops another condition, he/she is permitted on other clinical trials to treat that condition. Subjects are not permitted to go on other clinical trials for steroid refractory acute GVHD. Subjects are permitted to participate in trials for chronic GVHD.
* Pregnancy (a negative serum or urine pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation.
* Pre-existing or recent onset of demyelinating disorders
* Pre-existing or recent onset of gastrointestinal perforation
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to first infusion
* Previous treatment with Natalizumab (Tysabri®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Known active UNCONTROLLED bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds).
* Concomitant malignancies.
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* ANC < 0.5 x 103
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Serum creatinine > 1.9 mg/dL (168 µmol/L). Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times upper limit of normal (ULN) unless liver GVHD is suspected
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2014-06-17 (Actual); Study Completion 2014-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Usama Gergis, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Race (NIH/OMB)
Arm/Group | All Patients
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 60 [58 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With GVHD Who Are Tolerable to Tocilizumab After Having Failed Response to Glucocorticosteroid Treatment
Description: Both subjects enrolled on this study experienced failed response to glucocorticosteroid treatment but were able to tolerate tocilizumab. We were unable to collect extensive data on these 2 subjects because they both died early on in the study due to disease complications.
Time Frame: Day 28
Population: Not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 2
Participants | 2
Statistical Analysis 1: Comparison: All Patients; Not evaluable; Test type: Other — Not evaluable; Not evaluable; Other = 0; Not evaluable

2. Secondary Outcome: Disease-free Overall Survival at 100 Days, 6 Months and One Year From the Time of the First Tocilizumab Infusion.
Description: We were unable to evaluate disease-free survival at 100 days, 6 months and one year from the time of the first tocilizumab infusion. All subjects enrolled on this study died before this time point and the study closed to enrollment due to slow accrual.
Time Frame: Approximately 1 year
Population: We were unable to evaluate disease-free survival at 100 days, 6 months and one year from the time of the first tocilizumab infusion. All subjects enrolled on this study died before this time point and the study closed to enrollment due to slow accrual.
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Toclizumab Response in Each Organ
Description: We were unable to assess the Tocilizumab response in each organ at 1 year. All subjects enrolled on this study died before this time point and the study closed to enrollment due to slow accrual.
Time Frame: 1 year
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Effect of Toclizumab on Karnofsky Performance Status
Description: We were unable to evaluate the effect of tocilizumab on Karnofsky Performance Status at 1 year. All subjects enrolled on this study died before this time point and the study closed to enrollment due to slow accrual.
Time Frame: 1 year
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=2)
GVHD (Gastrointestinal disorders) | 1 (1) — gut GVHD grade 5
pulmonary infilatrates (Respiratory, thoracic and mediastinal disorders) | 1 — probably mycobacterium Kansasii

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No